CLINICAL TRIAL: NCT06058702
Title: Genetics of Cannabis Use Disorder and Cannabinoid Response in Humans
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Albert E. Kent Endowed Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2000036194; RO1 (Other: National Institute on Drug Abuse)
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Cannabis Use Disorder
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Delta-9-THC Very Low Dose (Active Comparator): Active delta-9-THC administered intravenously over 20 minutes.
  Interventions: Drug: Delta-9-THC Very Low Dose
- Placebo (Placebo Comparator): Control: small amount of alcohol administered intravenously (quarter teaspoon), with no delta-9-THC, over 20 minutes.
  Interventions: Drug: Placebo
- Delta-9-THC Medium Dose (Active Comparator): Active delta-9-THC administered intravenously over 20 minutes.
  Interventions: Drug: Delta-9-THC Medium Dose

INTERVENTIONS:
Drug: Delta-9-THC Very Low Dose — Active Delta-9-THC administered intravenously over 20 minutes.
  Arms: Delta-9-THC Very Low Dose
Drug: Placebo — Control: Small amount of sterile 190 proof USP ethanol (1-2 mLs), with no THC, administered intravenously over 20 minutes.
  Arms: Placebo
Drug: Delta-9-THC Medium Dose — Active Delta-9-THC administered intravenously over 20 minutes.
  Arms: Delta-9-THC Medium Dose

SUMMARY:
Cannabis is widely used worldwide and is associated with negative outcomes including cannabis use disorder (CanUD), psychosis, and cognitive impairment amongst others. Given the legalization of "recreational" and "medical" cannabis globally, the increasing availability of cannabis, the higher potency of cannabis, the availability of highly potent cannabinoid products, the commercialization of cannabis, and the rising rates of cannabis use, it is critical to understand how genetic factors influence 1) an individual's vulnerability for addiction and psychosis, 2) the response to cannabinoids, 3) the response to novel treatments for CanUD. CanUD is strongly genetically influenced; the investigators published the first CanUD genomewide association study (GWAS) with genomewide-significant results; however, the precise nature of the contribution of genetic factors in the development of CanUD is still not clear. Cannabis exposure has also been linked to a number of psychosis outcomes including schizophrenia (SCZ). SCZ is highly heritable and population-based and genetics studies both support a bidirectional genetic relationship between SCZ and CanUD. However, the precise contribution of genetic factors in the development of psychosis outcomes related to cannabis are not clear.

ELIGIBILITY:
Inclusion Criteria:

-Ages 21-60 years old

Exclusion Criteria:

* Major or unstable medical conditions based on history, the Structured Clinical Interview for DSM-5, collateral information, physical and laboratory examinations, ECG, and vital signs.
* Cannabis naïve individuals
* Positive pregnancy test

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 215 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Measured at baseline, 20 minutes, 45 minutes, 90 minutes, 140 minutes, 165 minutes, 210 minutes, 270 minutes, and 360 minutes after the start of the initial THC/placebo drug infusion.
  The VAS is a scale to document perceived reward. A higher score reflects a positive response.
Positive and Negative Symptom Scale (PANSS) | Measured at baseline, 45 minutes, 90 minutes, 165 minutes, 210 minutes, and 360 minutes after the start of the initial THC/placebo drug infusion.
  The Positive and Negative Syndrome Scale is a 30-item scale to assess both the positive and negative symptom symptoms of schizophrenia. The range total score is 30-210. An improvement in symptoms is reflected by a lower score.
Clinician Administered Dissociative Symptoms Scale (CADSS), | Measured at baseline, 45 minutes, 90 minutes, 165 minutes, 210 minutes, and 360 minutes after the start of the initial THC/placebo drug infusion.
  Perceptual alterations will be measured using scales such as the Clinician Administered Dissociative Symptoms Scale (CADSS), a scale consisting of 19 self-report items and 8 clinician-rated items (0 = not at all, 4 = extremely) that we have shown to be sensitive to THC effects. The scale captures alterations in environmental/time/body perception, feelings of unreality, and memory impairment.
CogState Battery | Measured at baseline, 45 minutes, and 165 minutes after the start of the initial THC/placebo drug infusion.
  The CogState Battery measures cognition including verbal learning and recall and episodic memory.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak D'Souza, MD, Principal Investigator — Yale University
Locations (1):
- West Haven Veterans Affairs Medical Center, West Haven, Connecticut, United States